CLINICAL TRIAL: NCT02734342
Title: Mixed Methods Study to Evaluate Pain, Function, Postural Stabilisation, and Fear of Movement Following a Lower Limb Exercise Programme for Knee Osteoarthritis
Brief Title: Mixed Methods Assessment of Exercises for Knee OA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Salford (Other)
Responsible Party: Principal Investigator, Jimmy Molyneux, Physiotherapist, University of Salford
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS ID 154227
Record Dates: First submitted 2016-02-15; First posted 2016-04-12 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise, Kinesiophobia and Knee Osteoarthritis (Experimental): Participants will be asked to attend eight exercise sessions within a group class environment that will last for 1 hour. During the hour, participants will complete a 5 minute warm up followed by 14 exercises specific to strengthening the lower limb and improve aerobic capacity. Each exercise will be timed for two minutes with the participant reporting number of repetitions counted.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — Participants will be asked to attend eight exercise sessions within a group class environment that will last for 1 hour. The exercise programme has been developed through clinical and research evidence. During the hour, a 5 minute warm up followed by 14 exercises specific to strengthening the lower limb and improving aerobic capacity. Each exercise will be timed for two minutes with the participant reporting number of repetitions counted. A cool down will be completed at the end of the class. After each exercise class, the participant will be advised to have a recovery day to prevent overloading (De Carlo & Armstrong, 2010). Progression of exercises will be patient led. Participants will attend twice per week for four weeks.

SUMMARY:
Osteoarthritis (OA) is a condition that causes cartilage loss, bony remodeling, joint stiffness and generalized muscle weakness. 90% of OA presentation has been reported within the leg; with 44% affecting the knee joint. Knee OA is expected to increase by 50% over the next twenty years due to an ageing population, obesity, and societal trends such as lack of activity. Only 13% of knee OA sufferers reach the recommended levels of exercise therefore an understanding of how psychological and functional relationships effect exercise engagement, which in turn would provide a more comprehensive rehabilitation programme for patients with knee OA. The aim of this study is to investigate exercise in knee OA and it it's correlation with fear of movement, using a mixed methods approach. Quantitative methodology will investigate lower limb exercises for pain and function and fear of movement. The desired outcome of the study will show that a reduction in pain with patient specific exercise will also reduce the fear of movement and allow patients to self-manage their symptoms without fear. Other quantitative factors such as intensity of exercise and postural stabilization using the Y balance test will also be utilized to review the functional relationship of muscle strength and balance to kinesiophobia. A semi-structured interview will be completed at the end of the course of treatment to highlight what patients think about exercise as an intervention. Participants aged forty-five and above with specific clinical symptoms will be invited into the study and will be asked to attend eight exercise sessions within a class environment, which will last for 1 hour within the Physiotherapy Department.

DETAILED DESCRIPTION:
Exercise is recommended for the treatment for knee osteoarthritis (OA) with muscle strength and aerobic exercise improving physical function. There is evidence supporting quadriceps strength for patients with painful knee OA; positive effects on pain; and general fitness.

Research reviews by suggest exercise as an important aspect of rehabilitation in knee OA. However, there is very limited evidence to what type of exercises actually decrease pain and improve activity.

Despite positive evidence regarding exercise, highlighted major issues within the United Kingdom with only 5% of people with knee OA achieving the recommended level of activity and 57% of the population not completing regular exercise. 1% to 4% of total healthcare costs account for physical inactivity which cost 8.3 billion in 2009.

An essential factor of physical inactivity is exercise behaviour. Fear of movement is an important aspect of knee OA. Disability is present due to the individual's fear of physical movements that would cause pain. Evidence links fear of movement with knee OA and the role of exercise in the management of knee OA. Patients with OA experience pain during activity, which leads to an expectation that further activity, will cause greater pain therefore increasing muscle weakness. It has been indicated that individuals could have negative attitudes and beliefs about their knee problems, which could cause a barrier to treatment, with socioeconomic, personality and environmental factors being as important as the physical characteristics. Other factors such as balance issues and laxity of the knee have been associated with activity limitations. However, in a systematic review found weak evidence to support pain, distress, and avoidance of activity in participants with knee OA. Understanding individual exercise behaviours and habits is essential to improve exercise adherence. Non-compliance is common within physiotherapy with patients unwilling to accommodate exercises within everyday life. Reasons for this may include type of exercises, dosage, and underlying beliefs from the clinicians towards exercise as well as external factors. Incorrect prescription of exercises can lead to increased pain, decreased function and decreased exercise adherence. This could cause fear of movement whilst completing exercise. It has been concluded that in OA there is limited evidence that interventions can improve exercise adherence. Therefore, an understanding of non-adherence and the effects of kinesiophobia is essential to further develop exercise programmes for patients with OA.

ELIGIBILITY:
Inclusion Criteria:

Patients must elicit 3 of the 6 symptoms to be included:

* forty five years of age and over.
* stiffness for less than thirty minutes;
* crepitus;
* bony tenderness;
* bony enlargement;
* no palpable joint warmth.

Exclusion Criteria:

* previous lower limb joint injection within three months;
* previous hip or knee joint replacement;
* any severe cognitive, cardio- respiratory, musculoskeletal or neurological - diagnosis that prevents participants from exercising;
* insoles or braces;
* ligament instability;
* participants with a body mass index (BMI) over 40 will be issued with a choice of completing in the study or being managed by the National Health Service weight management service;
* other minor health related issues will be assessed prior to the commencement of the study to ensure safe practice.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Change in the level of kinesiophobia with exercise assessed using the Tampa Kinesiophobia Scale during an exercise programme and 6 weeks after the programme. | At the beginning, through study completion, an average 10 weeks.
  Patients will be asked to complete the Tampa Kinesiophobia Scale at the beginning of the study, before exercise session 4, before session 8 and 6 weeks after the exercise programme. This will measure the level of kinesiophobia associated with exercise. If an individual scores highly, this indicates a high level of kinesiophobia.

SECONDARY OUTCOMES:
Change in the level of psychological and functional relationships using the Y balance test during an exercises programme and 6 weeks after the programme. | At the beginning, through study completion, an average 10 weeks.
  The Y balance test is a quick, efficient, objective, portable, and consistent tool and will be used to evaluate dynamic and asymmetrical balance whilst utilising muscle strength and flexibility at the hip, knee and ankle joints. It consists of a stance platform to which three pieces of plastic pipe are attached in the three reach directions; anterior (ANT), posteromedial (PM), and posterolateral (PL). The PM and PL pipes are positioned 135 degrees from the ANT pipe with 45 degrees between the posterior pipes. The pipes are marked at 5 mm intervals for measurement. To perform the test the subject pushes the reach indicator along each of the pipes and a score is calculated. Each leg will be tested.
Change in the understanding of key factors that patients think about exercise as an intervention using a semistructured interview. | 6 weeks post exercise class
  A semi-structured interview will be completed at the end of course of treatment to highlight what patients think about exercise as an intervention.

OTHER OUTCOMES:
Change in the level of function, pain,quality of life, sport and recreation, activities of daily living and symptoms in patients during an exercise programme and 6 weeks after the programme. | At the beginning, through study completion, an average 10 weeks.
  Knee injury and Osteoarthritis Outcome Score (KOOS) is a valid, highly reliable, and responsive for evaluating changes after OA interventions. This is a questionnaire that consists of 42 questions covering Pain; Symptoms; Function in Daily Living Function in Sport and Recreation and Knee-Related Quality of Life. The score is then normalized to a 0-100 scale with the higher score being better.
Change in the level of physical activity during an exercise programme and 6 weeks after the programme. | At the beginning, through study completion, an average 10 weeks.
  Physical activity will be measured using the physical activity scale for the elderly (PASE), which is a valid and reliable measurement tool. It is a self-administered questionnaire, which assesses a wide range of activities such as leisure time activity, household activity, and work related activity. It consists of 12 questions and is calculated by multiplying either the time spent in each activity (hours per week) or participation in an activity. The overall scores ranges' from 0-400.
Change in the distance walked within a 6 minute period during an exercise programme and 6 weeks after the programme. | At the beginning, through study completion, an average 10 weeks.
  A 6 minute walk test to assess aerobic walking capacity; dynamic balance whilst changing direction and maximal distance covered in a 6-minute period.
Change in the level of pain intensity during an exercise programme and 6 weeks after the programme. | At the beginning, through study completion, an average 10 weeks.
  Visual Analogue Scale (VAS) is an horizontal line, 100 mm in length, anchored by word descriptors at each end. The patient marks on the line the point that they feel represents their perception of their current pain intensity. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.
Change in the level of perceived exertion during an exercise programme . | At the beginning, through study completion, an average 4 weeks.
  Modified Borg scale for exercise intensity tool will be used. It will be used to document the patient's exertion after the exercise programme and is used to assess the intensity of training. The exertion is rated on a scale of 6-20, where 6 means "no exertion at all" and 20 means "maximal exertion.
Change in the level of physical activity during an exercise programme and 6 weeks after the programme. | At the beginning and 6 weeks after the exercise programme.
  An activity monitor will be issued to monitor physical activity and should be worn continuously for 7 days during waking hours. The Activity monitor is a device that measures the postural aspect of inactivity. It is a small monitor that is placed on the midline anterior aspect of the upper thigh and can determine body position, such as sitting, lying, being upright and movements between these postures, stepping and stepping speed.
Change in the level of lower extremity functional strength during an exercise programme and 6 weeks after the programme. | At the beginning, through study completion, an average 10 weeks.
  The 30 second chair test is administered using a folding chair without arms, with seat height of 17 inches (43.2 cm). The chair, with rubber tips on the legs, is placed against a wall to prevent it from moving.
  The participant is seated in the middle of the chair, back straight; feet approximately shoulder width apart and placed on the floor at an angle slightly back from the knees, with one foot slightly in front of the other to help maintain balance. Arms are crossed at the wrists and held against the chest. The participant is encouraged to complete as many full stands as possible within 30 seconds. The participant is instructed to fully sit between each stand.The 30 second chair stand involves recording the number of stands a person can complete in 30 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Bridgewater Community Healthcare Foundation Trust, Leigh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The results of the study will form part of the researcher's doctoral thesis and may be published anonymously in professional journals and/or as conference presentations.

REFERENCES:
- [Derived] Molyneux J, Herrrington L, Riley B, Jones R. A single-arm, non-randomized investigation into the short-term effects and follow-up of a 4-week lower limb exercise programme on kinesiophobia in individuals with knee osteoarthritis. Physiother Res Int. 2020 Jul;25(3):e1831. doi: 10.1002/pri.1831. Epub 2020 Jan 24. PMID 31975503